CLINICAL TRIAL: NCT04729452
Title: Characterisation of the Immune Response to SARS-CoV-2 Infection
Brief Title: Characterisation of the Immune Response to SARS-CoV-2 / COVID-19
Status: Completed | Type: Observational
Sponsor: Cwm Taf University Health Board (NHS) (Other Government)
Collaborators: Cardiff University (Other); University of Oxford (Other)
Responsible Party: Principal Investigator, Lucy Jones, Honorary Clinical Lecturer and Associate Specialist, Cwm Taf University Health Board (NHS)
Other Study IDs: CT 269506
Record Dates: First submitted 2021-01-25; First posted 2021-01-28 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: blood test — blood test to test immune response to SARS-CoV-2
  Other Names: serial blood tests over 6 months

SUMMARY:
Emerging clinical details of the current SARS-CoV-2 pandemic have illustrated that there are multiple clinical presentations and outcomes of this viral infection. People with an infection have been reported to have a spectrum of disease from severe acute respiratory distress requiring ventilation, to mild respiratory or gastrointestinal symptoms and asymptomatic presentations. Mechanisms explaining the heterogeneity of host response to infection are yet to be characterised.

The aim of this project is to understand the host immune response to infection with SARS-CoV-2 over time in convalescent adults, including acquired immune responses, circulating levels of immune signalling molecules, gene expression profiling in peripheral blood and to identify host genetic variants associated with disease progressions or severity. Participants will be healthcare workers who had a diagnosis of COVID-19 (confirmed by positive RT-PCR assay) more than 28 days ago and have recovered and are employed by Cwm Taf Morgannwg University health board. Samples will be processed and analysed to explore immunological, host genetic factors and virological factors that explain pathogenesis and predict outcomes of infection.

DETAILED DESCRIPTION:
AIMS AND OBJECTIVES The objective of this project is to understand the host immune response to infection with SARS-CoV-2 over time in convalescent adults, including acquired immune responses, gene expression profiling in peripheral blood and to identify host genetic variants associated with disease progressions or severity. We would like to ascertain why different people experience different disease phenotypes with this coronavirus infection.

Our primary objective is to determine key protective cellular immune parameters (e.g. T cell responses) and confirm whether there are host genetic factors that provide protection from disease. We aim to define immunodominant SARS-CoV-2 T-cell epitopes by screening overlapping peptides from the viral proteome and mapping responses to individual COVID proteins expressed intracellularly in antigen-presenting cells (to confirm processing and presentation at the cell surface). Peptide-HLA multimers will be constructed for confirmed immunodominant responses. These reagents will allow rapid enumeration and tracking of COVID-specific T cell responses in patient samples.

Our secondary objective is to determine whether there are public (shared) T-cell receptor responses to SARS-CoV-2. We will also examine whether pre-existing T-cells responses to other viruses protect against SARS-CoV-2-induced disease (COVID-19). T-cells generated will be used to test and verify detection reagents. These reagents will be developed for various projects in Oxford University including monitoring of T-cell responses induced by COVID vaccines. We will also establish whether pre-existing cross-reactive immunity to other coronaviruses correlates with disease severity as seen with the 2009 swine flu pandemic.

ELIGIBILITY:
Inclusion Criteria:

The study will enrol eligible participants with confirmed COVID-19 PCR-based test 28 or more days prior to recruitment and be convalescent. Participants must be 18 years old and must have the capacity to provide written consent after discussing the participant information sheet. Participants must be health care workers for Cwm Taf Morgannwg University Health board.

Exclusion Criteria:

Participants who are acutely unwell with COVID. Participants who cannot provide informed written consent. Participants who have a clear co-infection with a relevant pathogen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health care workers who had a positive SARS-CoV-2 nasopharyngeal swab test more than 28 days before recruitment
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Determination of key protective cellular immune parameters | 2 years
  Our primary objective is to determine key protective cellular immune parameters (e.g. T cell responses) and confirm whether there are host genetic factors that provide protection from disease. We aim to define immunodominant SARS-CoV-2 T-cell epitopes by screening overlapping peptides from the viral proteome and mapping responses to individual COVID proteins expressed intracellularly in antigen-presenting cells (to confirm processing and presentation at the cell surface). Peptide-HLA multimers will be constructed for confirmed immunodominant responses. These reagents will allow rapid enumeration and tracking of COVID-specific T cell responses in patient samples.

SECONDARY OUTCOMES:
Determination of public T-cell receptor response to SARS-CoV-2 | 3 years
  Our secondary objective is to determine whether there are public (shared) T-cell receptor responses to SARS-CoV-2. We will also examine whether pre-existing T-cells responses to other viruses protect against SARS-CoV-2-induced disease (COVID-19). T-cells generated will be used to test and verify detection reagents. These reagents will be developed for various projects in Oxford University including monitoring of T-cell responses induced by COVID vaccines. We will also establish whether pre-existing cross-reactive immunity to other coronaviruses correlates with disease severity as seen with the 2009 swine flu pandemic.

CONTACTS AND LOCATIONS:
Locations (1):
- Cwm Taf Morgannwg University Health board, Llantrisant, Rhondda Cynon Taf, United Kingdom

IPD SHARING:
Plan to Share IPD: No